CLINICAL TRIAL: NCT03484429
Title: Effects of Postoperative Percutaneous Peripheral Nerve Stimulation on Acute and Chronic Amputation Pain
Brief Title: Postoperative Peripheral Nerve Stimulation for Management of Post-amputation Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2343
Record Dates: First submitted 2018-02-07; First posted 2018-03-30 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Phantom Limb Pain; Postoperative Pain; Neuroma; Acute Pain; Chronic Pain; Residual Limbs; Amputation
Keywords: Neurostimulation; Peripheral nerve stimulation
MeSH Terms: conditions — Phantom Limb; Pain, Postoperative; Neuroma; Acute Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Experimental): Standard medical therapy and 30 to 60 days of peripheral nerve stimulation starting within 7 days after surgery
  Interventions: Device: Peripheral nerve stimulation; Other: Standard Medical Therapy
- Group 2 (Active Comparator): Standard medical therapy only
  Interventions: Other: Standard Medical Therapy

INTERVENTIONS:
Device: Peripheral nerve stimulation — Up to 60 days of peripheral nerve stimulation
  Arms: Group 1
Other: Standard Medical Therapy — Medications, physical therapy, or other pain treatments

SUMMARY:
Limb loss is frequently associated with postamputation pain that can be challenging to treat and often involves opioids. Advances in the field of neuromodulation has led to development of an intentionally reversible percutaneous peripheral nerve stimulation (PNS) system that has had promising results when treating chronic postamputation pain. PNS may offer sustained pain relief even after the treatment period has ended. Currently, there is no convincing evidence regarding the role of PNS in the acute postoperative period, which may be a critical time to control pain as those with higher pain appear to be at higher risk for developing persistent post-procedural pain. The investigators of this study aim to evaluate the feasibility and effects of PNS in the acute postoperative period and determine the feasibility of completing a randomized controlled treatment outcome study.

DETAILED DESCRIPTION:
16 patients with new nontraumatic transfemoral or transtibial amputation will be enrolled in the study

Having met inclusion criteria, the patients will be randomized to experimental or control groups

Patients in the experimental group undergo placement of PNS leads within 7 days of amputation surgery

Patients in both groups will be treated with standard pharmacologic and nonpharmacologic pain therapies and evaluated weekly for 8 weeks, then at 3, 6, and 12 months postamputation

ELIGIBILITY:
Inclusion Criteria:

* Nontraumatic transfemoral (above-the-knee) or transtibial (below-the-knee) amputation
* Presence of postamputation pain rated at least 4 or more

Exclusion Criteria:

* Beck Depression Inventory score greater than 20
* Systemic infection
* Immunocompromised or taking immunosuppressive medications
* Implanted electronic device
* Pregnancy
* Previous allergy to skin contact materials and/or anesthetic agent
* Altered mental status
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Lester, MD, Principal Investigator — Hunter Holmes McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hanley MA, Jensen MP, Smith DG, Ehde DM, Edwards WT, Robinson LR. Preamputation pain and acute pain predict chronic pain after lower extremity amputation. J Pain. 2007 Feb;8(2):102-9. doi: 10.1016/j.jpain.2006.06.004. Epub 2006 Sep 1. PMID 16949876
- [Background] Karanikolas M, Aretha D, Tsolakis I, Monantera G, Kiekkas P, Papadoulas S, Swarm RA, Filos KS. Optimized perioperative analgesia reduces chronic phantom limb pain intensity, prevalence, and frequency: a prospective, randomized, clinical trial. Anesthesiology. 2011 May;114(5):1144-54. doi: 10.1097/ALN.0b013e31820fc7d2. PMID 21368651
- [Background] Kent ML, Hsia HJ, Van de Ven TJ, Buchheit TE. Perioperative Pain Management Strategies for Amputation: A Topical Review. Pain Med. 2017 Mar 1;18(3):504-519. doi: 10.1093/pm/pnw110. PMID 27402960
- [Background] Capdevila X, Bringuier S, Borgeat A. Infectious risk of continuous peripheral nerve blocks. Anesthesiology. 2009 Jan;110(1):182-8. doi: 10.1097/ALN.0b013e318190bd5b. No abstract available. PMID 19104185
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Ilfeld BM, Grant SA. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation for Postoperative Analgesia: Could Neurostimulation Replace Continuous Peripheral Nerve Blocks? Reg Anesth Pain Med. 2016 Nov/Dec;41(6):720-722. doi: 10.1097/AAP.0000000000000481. No abstract available. PMID 27685345
- [Background] Ilfeld BM, Gabriel RA, Saulino MF, Chae J, Peckham PH, Grant SA, Gilmore CA, Donohue MC, deBock MG, Wongsarnpigoon A, Boggs JW. Infection Rates of Electrical Leads Used for Percutaneous Neurostimulation of the Peripheral Nervous System. Pain Pract. 2017 Jul;17(6):753-762. doi: 10.1111/papr.12523. Epub 2016 Nov 11. PMID 27676323
- [Background] Ilfeld BM, Ball ST, Gabriel RA, Sztain JF, Monahan AM, Abramson WB, Khatibi B, Said ET, Parekh J, Grant SA, Wongsarnpigoon A, Boggs JW. A Feasibility Study of Percutaneous Peripheral Nerve Stimulation for the Treatment of Postoperative Pain Following Total Knee Arthroplasty. Neuromodulation. 2019 Jul;22(5):653-660. doi: 10.1111/ner.12790. Epub 2018 Jul 19. PMID 30024078
- [Background] Ilfeld BM, Gabriel RA, Said ET, Monahan AM, Sztain JF, Abramson WB, Khatibi B, Finneran JJ 4th, Jaeger PT, Schwartz AK, Ahmed SS. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Sciatic Nerve for Postoperative Analgesia Following Ambulatory Foot Surgery, a Proof-of-Concept Study. Reg Anesth Pain Med. 2018 Aug;43(6):580-589. doi: 10.1097/AAP.0000000000000819. PMID 29905630
- [Background] Ilfeld BM, Finneran JJ 4th, Gabriel RA, Said ET, Nguyen PL, Abramson WB, Khatibi B, Sztain JF, Swisher MW, Jaeger P, Covey DC, Meunier MJ, Hentzen ER, Robertson CM. Ultrasound-guided percutaneous peripheral nerve stimulation: neuromodulation of the suprascapular nerve and brachial plexus for postoperative analgesia following ambulatory rotator cuff repair. A proof-of-concept study. Reg Anesth Pain Med. 2019 Mar;44(3):310-318. doi: 10.1136/rapm-2018-100121. Epub 2019 Feb 15. PMID 30770421
- [Background] Gilmore C, Ilfeld B, Rosenow J, Li S, Desai M, Hunter C, Rauck R, Kapural L, Nader A, Mak J, Cohen S, Crosby N, Boggs J. Percutaneous peripheral nerve stimulation for the treatment of chronic neuropathic postamputation pain: a multicenter, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2019 Jun;44(6):637-645. doi: 10.1136/rapm-2018-100109. Epub 2019 Apr 5. PMID 30954936
- [Background] Gilmore CA, Ilfeld BM, Rosenow JM, Li S, Desai MJ, Hunter CW, Rauck RL, Nader A, Mak J, Cohen SP, Crosby ND, Boggs JW. Percutaneous 60-day peripheral nerve stimulation implant provides sustained relief of chronic pain following amputation: 12-month follow-up of a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2019 Nov 17:rapm-2019-100937. doi: 10.1136/rapm-2019-100937. Online ahead of print. PMID 31740443
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Linacre JM, Heinemann AW, Wright BD, Granger CV, Hamilton BB. The structure and stability of the Functional Independence Measure. Arch Phys Med Rehabil. 1994 Feb;75(2):127-32. PMID 8311667
- [Background] Anagnostis C, Gatchel RJ, Mayer TG. The pain disability questionnaire: a new psychometrically sound measure for chronic musculoskeletal disorders. Spine (Phila Pa 1976). 2004 Oct 15;29(20):2290-302; discussion 2303. doi: 10.1097/01.brs.0000142221.88111.0f. PMID 15480144
- [Background] Massarweh NN, Kaji AH, Itani KMF. Practical Guide to Surgical Data Sets: Veterans Affairs Surgical Quality Improvement Program (VASQIP). JAMA Surg. 2018 Aug 1;153(8):768-769. doi: 10.1001/jamasurg.2018.0504. No abstract available. PMID 29617543
- [Background] Deer TR, Mekhail N, Provenzano D, Pope J, Krames E, Leong M, Levy RM, Abejon D, Buchser E, Burton A, Buvanendran A, Candido K, Caraway D, Cousins M, DeJongste M, Diwan S, Eldabe S, Gatzinsky K, Foreman RD, Hayek S, Kim P, Kinfe T, Kloth D, Kumar K, Rizvi S, Lad SP, Liem L, Linderoth B, Mackey S, McDowell G, McRoberts P, Poree L, Prager J, Raso L, Rauck R, Russo M, Simpson B, Slavin K, Staats P, Stanton-Hicks M, Verrills P, Wellington J, Williams K, North R; Neuromodulation Appropriateness Consensus Committee. The appropriate use of neurostimulation of the spinal cord and peripheral nervous system for the treatment of chronic pain and ischemic diseases: the Neuromodulation Appropriateness Consensus Committee. Neuromodulation. 2014 Aug;17(6):515-50; discussion 550. doi: 10.1111/ner.12208. PMID 25112889
- [Background] Deer TR, Naidu R, Strand N, Sparks D, Abd-Elsayed A, Kalia H, Hah JM, Mehta P, Sayed D, Gulati A. A review of the bioelectronic implications of stimulation of the peripheral nervous system for chronic pain conditions. Bioelectron Med. 2020 Apr 24;6:9. doi: 10.1186/s42234-020-00045-5. eCollection 2020. PMID 32346553
- [Background] Rauck RL, Cohen SP, Gilmore CA, North JM, Kapural L, Zang RH, Grill JH, Boggs JW. Treatment of post-amputation pain with peripheral nerve stimulation. Neuromodulation. 2014 Feb;17(2):188-97. doi: 10.1111/ner.12102. Epub 2013 Aug 15. PMID 23947830
- [Background] Bruce J, Quinlan J. Chronic Post Surgical Pain. Rev Pain. 2011 Sep;5(3):23-9. doi: 10.1177/204946371100500306. PMID 26526062
- [Background] Imani F. Postoperative pain management. Anesth Pain Med. 2011 Jul;1(1):6-7. doi: 10.5812/kowsar.22287523.1810. Epub 2011 Jul 1. No abstract available. PMID 25729647
- [Background] Borghi B, D'Addabbo M, White PF, Gallerani P, Toccaceli L, Raffaeli W, Tognu A, Fabbri N, Mercuri M. The use of prolonged peripheral neural blockade after lower extremity amputation: the effect on symptoms associated with phantom limb syndrome. Anesth Analg. 2010 Nov;111(5):1308-15. doi: 10.1213/ANE.0b013e3181f4e848. Epub 2010 Sep 29. PMID 20881281
- [Background] Columbo JA, Davies L, Kang R, Barnes JA, Leinweber KA, Suckow BD, Goodney PP, Stone DH. Patient Experience of Recovery After Major Leg Amputation for Arterial Disease. Vasc Endovascular Surg. 2018 May;52(4):262-268. doi: 10.1177/1538574418761984. Epub 2018 Mar 1. PMID 29495957
- [Background] Houghton AD, Nicholls G, Houghton AL, Saadah E, McColl L. Phantom pain: natural history and association with rehabilitation. Ann R Coll Surg Engl. 1994 Jan;76(1):22-5. PMID 8117013
- [Background] Gallagher P, Allen D, Maclachlan M. Phantom limb pain and residual limb pain following lower limb amputation: a descriptive analysis. Disabil Rehabil. 2001 Aug 15;23(12):522-30. doi: 10.1080/09638280010029859. PMID 11432649
- [Background] Raichle KA, Hanley MA, Molton I, Kadel NJ, Campbell K, Phelps E, Ehde D, Smith DG. Prosthesis use in persons with lower- and upper-limb amputation. J Rehabil Res Dev. 2008;45(7):961-72. doi: 10.1682/jrrd.2007.09.0151. PMID 19165686
- [Background] Armaghani SJ, Lee DS, Bible JE, Archer KR, Shau DN, Kay H, Zhang C, McGirt MJ, Devin CJ. Preoperative opioid use and its association with perioperative opioid demand and postoperative opioid independence in patients undergoing spine surgery. Spine (Phila Pa 1976). 2014 Dec 1;39(25):E1524-30. doi: 10.1097/BRS.0000000000000622. PMID 25417827
- [Background] Smith SR, Bido J, Collins JE, Yang H, Katz JN, Losina E. Impact of Preoperative Opioid Use on Total Knee Arthroplasty Outcomes. J Bone Joint Surg Am. 2017 May 17;99(10):803-808. doi: 10.2106/JBJS.16.01200. PMID 28509820
- [Derived] Albright-Trainer B, Phan T, Trainer RJ, Crosby ND, Murphy DP, Disalvo P, Amendola M, Lester DD. Peripheral nerve stimulation for the management of acute and subacute post-amputation pain: a randomized, controlled feasibility trial. Pain Manag. 2022 Apr;12(3):357-369. doi: 10.2217/pmt-2021-0087. Epub 2021 Nov 11. PMID 34761694

RESULTS

PARTICIPANT FLOW:
Groups:
- Peripheral Nerve Stimulation (PNS): Standard medical therapy and 30 to 60 days of peripheral nerve stimulation starting within 7 days after surgery
  Peripheral nerve stimulation: Up to 60 days of peripheral nerve stimulation
  Standard Medical Therapy: Medications, physical therapy, or other pain treatments
- Standard Medical Therapy (SMT): Standard medical therapy only
  Standard Medical Therapy: Medications, physical therapy, or other pain treatments
Period: Overall Study
Arm/Group | Peripheral Nerve Stimulation (PNS) | Standard Medical Therapy (SMT)
Started | 8 | 8
Postamputation Week 1-4 | 8 | 8
Postamputation Week 5-8 | 5 | 8
Postamputation Month 3 | 5 | 7
Completed | 5 | 8
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Peripheral Nerve Stimulation (PNS): Up to 60 days of PNS starting within 7 days after major lower limb amputation surgery. Subjects also received standard medical therapy (SMT). SMT is defined as pharmacotherapy, physical therapy, or other therapies.
- Control: Subjects received SMT only after major lower limb amputation surgery. SMT is defined as pharmacotherapy, physical therapy, or other therapies.
- Total: Total of all reporting groups
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Perineural Catheter Infusion [Mean (Standard Deviation); unit: Days] | 6 (1) | 5.5 (2.5) | 5.75 (2.5)
Taking Opioids Preoperatively [Count of Participants; unit: Participants] | 3 | 2 | 5
Level of Amputation [Count of Participants; unit: Participants]
  Above Knee | 5 | 4 | 9
  Below Knee | 3 | 4 | 7
Indication for Surgery [Count of Participants; unit: Participants]
  Peripheral Vascular Disease (PVD) | 3 | 4 | 7
  Peripheral Arterial Disease (PAD) | 2 | 1 | 3
  Pain | 2 | 0 | 2
  Diabetes (DM) | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Phantom Limb Pain (PLP) Score
Description: Using the Brief Pain Inventory-Short Form (BPI-SF) questionnaire, subjects were asked to rate their PLP over the past 24 hours on a scale of "0"=no pain to "10"=worst pain they have ever experienced. A lower score is better. Data from Weeks 1-4 and Weeks 5-8 were averaged to obtain a numerical score for these time points.
Time Frame: Baseline, Weeks 1-4, Weeks 5-8, and Month 3.
Population: Subjects who completed up to 60 days of peripheral nerve stimulation (PNS) and standard medical therapy (SMT) or (SMT) only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 4.1 (3.2) | 3.1 (2.7)
  Weeks 1-4 | 2.2 (2.4) | 3.0 (1.7)
  Weeks 5-8: number analyzed (Participants) | 5 | 8
  Weeks 5-8 | 1.0 (1.2) | 2.2 (2.2)
  Month 3: number analyzed (Participants) | 5 | 7
  Month 3 | 1.0 (1.2) | 1.3 (2.2)

2. Primary Outcome: Average Residual Limb Pain (RLP) Score
Description: Using the Brief Pain Inventory-Short Form (BPI-SF) questionnaire, subjects were asked to rate their RLP over the past 24 hours on a scale of "0"=no pain to "10"=worst pain they have ever experienced. A lower score is better. Data from Weeks 1-4 and Weeks 5-8 were averaged to obtain a numerical score for these time points.
Time Frame: Baseline, Weeks 1-4, Weeks 5-8, and Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 7.1 (2.2) | 4.4 (1.4)
  Weeks 1-4: number analyzed (Participants) | 5 | 8
  Weeks 1-4 | 3.6 (2.5) | 2.2 (1.6)
  Weeks 5-8: number analyzed (Participants) | 5 | 8
  Weeks 5-8 | 1 (1) | 2.1 (2)
  Month 3: number analyzed (Participants) | 5 | 7
  Month 3 | 0 (0) | 1.1 (1.9)

3. Primary Outcome: Worst Phantom Limb Pain (PLP) Score
Description: as for outcome 1
Time Frame: Baseline, Weeks 1-4, 5-8, and Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 6.5 (4.4) | 5.9 (4.0)
  Weeks 1-4 | 3.1 (3.1) | 5.4 (2.6)
  Weeks 5-8: number analyzed (Participants) | 5 | 8
  Weeks 5-8 | 2.2 (1.6) | 3.6 (3.3)
  Month 3: number analyzed (Participants) | 5 | 7
  Month 3 | 2.2 (2.7) | 2.0 (3.2)

4. Primary Outcome: Worst Residual Limb Pain (RLP) Score
Description: as for outcome 2
Time Frame: Baseline, Weeks 1-4, Weeks 5-8, and Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 8.3 (1.9) | 7.8 (1.9)
  Weeks 1-4 | 5.1 (2.6) | 4.1 (2.5)
  Weeks 5-8: number analyzed (Participants) | 5 | 8
  Weeks 5-8 | 1.7 (1.5) | 3.2 (2.7)
  Month 3: number analyzed (Participants) | 5 | 7
  Month 3 | 0 (0) | 1.9 (2.9)

5. Primary Outcome: Best Phantom Limb Pain (PLP) Score
Description: as for outcome 1
Time Frame: Baseline, Weeks 1-4, Weeks 5-8, and Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 1.4 (2.1) | 1.3 (1.6)
  Weeks 1-4 | 0.8 (1.1) | 1.4 (1.4)
  Weeks 5-8: number analyzed (Participants) | 5 | 8
  Weeks 5-8 | 0.6 (1.0) | 1.1 (0.9)
  Month 3: number analyzed (Participants) | 5 | 7
  Month 3 | 0.4 (0.7) | 1.0 (1.4)

6. Primary Outcome: Best Residual Limb Pain (RLP) Score
Description: as for outcome 2
Time Frame: Baseline, Weeks 1-4, Weeks 5-8, and Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline | 4.1 (2.6) | 1.5 (1.5)
  Weeks 1-4 | 1.7 (1.4) | 1.0 (0.8)
  Weeks 5-8: number analyzed (Participants) | 5 | 8
  Weeks 5-8 | 0.4 (0.7) | 1.0 (0.9)
  Month 3: number analyzed (Participants) | 5 | 7
  Month 3 | 0.0 (0.0) | 0.4 (1.1)

7. Secondary Outcome: Number Taking Opioids
Description: The number of subjects prescribed any opioid medication and any dose. Data from Weeks 1-4 and Weeks 5-8 were averaged to obtain a numerical score for these time points.
Time Frame: Preop, Hospital Discharge, Weeks 1-4, Weeks 5-8, Week 12
Population: Between Weeks 1-4 and Weeks 5-8, three subjects in the PNS Group terminated due to unrelated medical events (2) or withdrew consent (1). After Week 12, two subjects in the Control Group terminated due to unrelated medical events or withdrew consent (data for one subject was collected prior to withdrawal).
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
Participants
  Baseline | 3 | 2
  Hospital Discharge | 6 | 7
  Weeks 1-4 | 3 | 5
  Weeks 5-8: number analyzed (Participants) | 5 | 8
  Weeks 5-8 | 1 | 4
  Week 12: number analyzed (Participants) | 5 | 7
  Week 12 | 1 | 3

8. Secondary Outcome: Average Oral Morphine Equivalents (OME)
Description: Opioid consumption (daily OME) over time was collected for all subjects.
Time Frame: Preoperative, Hospital discharge, Weeks 1-4, Weeks 5-8, and Week 12
Population: All study participants were evaluated.
Measure: Mean (Standard Deviation); unit: oral morphine equivalents (mg)
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
oral morphine equivalents (mg)
  Preop | 36.1 (60.5) | 7.2 (13.3)
  Hospital Discharge | 44.1 (57.2) | 36.1 (30.4)
  Weeks 1-4 | 23.4 (47.7) | 16.6 (30.0)
  Weeks 5-8: number analyzed (Participants) | 5 | 8
  Weeks 5-8 | 13.5 (24.9) | 20.3 (31.0)
  Week 12: number analyzed (Participants) | 5 | 7
  Week 12 | 13.5 (23.9) | 10.7 (20.7)

9. Secondary Outcome: Functional Independence Measure (FIM) Scores
Description: FIM mobility subscores were recorded by a physical therapist to measure the ability to walk, use a wheelchair, transfer to tub/shower, transfer to toilet, and mobility in bed, chair, and wheelchair. Scores range from "1" = subject requires total assistance for the task to "7" = complete independence. A higher score is better.
Time Frame: Preoperative, Week 4, and Week 8
Population: All qualifying subjects were evaluated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Walk (Preop) | 1 (0) | 1 (0)
  Walk (Week 4): number analyzed (Participants) | 6 | 5
  Walk (Week 4) | 1 (0) | 1.2 (0.4)
  Walk (Week 8): number analyzed (Participants) | 7 | 7
  Walk (Week 8) | 1.7 (1.5) | 1.3 (0.8)
  Wheelchair (Preop) | 4.8 (1.6) | 5.4 (0.7)
  Wheelchair (Week 4): number analyzed (Participants) | 6 | 5
  Wheelchair (Week 4) | 5.8 (0.4) | 5.8 (0.4)
  Wheelchair (Week 8): number analyzed (Participants) | 7 | 7
  Wheelchair (Week 8) | 5.9 (0.4) | 6.1 (0.0)
  Tub/Shower Transfer (Preop) | 4.1 (1.6) | 4.1 (1.1)
  Tub/Shower Transfer (Week 4): number analyzed (Participants) | 6 | 5
  Tub/Shower Transfer (Week 4) | 5.8 (0.4) | 5.4 (1.5)
  Tub/Shower Transfer (Week 8): number analyzed (Participants) | 7 | 7
  Tub/Shower Transfer (Week 8) | 5.7 (0.5) | 5.7 (0.5)
  Toilet Transfer (Preop) | 4.6 (0.9) | 3.9 (1.4)
  Toilet Transfer (Week 4): number analyzed (Participants) | 6 | 5
  Toilet Transfer (Week 4) | 5.8 (0.4) | 5.0 (1.7)
  Toilet Transfer (Week 8): number analyzed (Participants) | 7 | 7
  Toilet Transfer (Week 8) | 5.7 (0.5) | 5.7 (0.5)
  Bed/Chair/Wheelchair Mobility (Preop) | 4.9 (1.0) | 4.3 (0.7)
  Bed/Chair/Wheelchair Mobility (Week 4) | 5.9 (0.4) | 5.7 (0.9)
  Bed/Chair/Wheelchair Mobility (Week 8) | 5.7 (0.5) | 6.0 (0.0)

10. Secondary Outcome: Pain Interference
Description: Using the Brief Pain Inventory-Short Form (BPI-SF) questionnaire, subjects were asked to rate how much pain has interfered with daily activities over the past 24 hours on a scale of "0" = no interference to "10" = completely interferes with activities. A lower score is better.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: Subjects who were enrolled in the study and for whom this data was collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 4 | 8
score on a scale
  Baseline: number analyzed (Participants) | 4 | 5
  Baseline | 2.7 (3.1) | 3.7 (2.3)
  Week 4 | 2 (2.6) | 1.1 (1.5)
  Week 8: number analyzed (Participants) | 4 | 5
  Week 8 | 1.0 (1.1) | 1.0 (2.1)
  Week 12: number analyzed (Participants) | 4 | 5
  Week 12 | 0.2 (0.4) | 0.8 (1.2)

11. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Self-report measure PGIC reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as
  1 = "very much improved," 2 = "much improved," 3 = "minimally improved," 4 = "no change," 5 = "minimally worse," 6 = "much worse," or 7 = "very much worse." A lower score is better.
Time Frame: Weeks 4, 8, and 12
Population: Subjects who were enrolled in the study and for whom this data was collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 7 | 8
score on a scale
  Week 4 | 4.3 (2.6) | 3.9 (2.2)
  Week 8 | 4.1 (2.7) | 5.1 (2.1)
  Week 12: number analyzed (Participants) | 5 | 7
  Week 12 | 3.8 (2.2) | 2.4 (1.5)

12. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: Pain catastrophizing is the tendency to magnify the threat value of a pain stimulus and to feel helpless in the presence of pain. This is further characterized by the inability to prevent or inhibit pain-related thoughts surrounding a painful event. Pain catastrophizing affects how individuals experience pain. The PCS is a 13-item inventory of statements in which the subject is asked to rate the degree to which they agree, on a scale of "0" = not at all to "4" = all the time. The responses for each item are added for a total PCS score (range 0-52). A lower score is better.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: Subjects who were enrolled in the study and for whom this data was collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline: number analyzed (Participants) | 8 | 6
  Baseline | 20.3 (7.7) | 12.3 (9.2)
  Week 4: number analyzed (Participants) | 4 | 7
  Week 4 | 10.3 (7.2) | 8 (10.4)
  Week 8: number analyzed (Participants) | 7 | 8
  Week 8 | 4.1 (10.1) | 4.6 (7.4)
  Week 12: number analyzed (Participants) | 3 | 6
  Week 12 | 17 (21.8) | 9.8 (14.3)

13. Secondary Outcome: Pain Disability Index (PDI)
Description: The PDI is designed to measure the degree to which aspects of life are disrupted by chronic pain. The impact of pain on various aspects of life (e.g. family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activities) are recorded on a 10-point scale from "0" = no disability to "10" = worst disability. The sum of scores is recorded for a total PDI score (range 0-70). A lower score is better.
Time Frame: Weeks 4, Week 8, and Week 12
Population: Subjects who were enrolled in the study and for whom this data was collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 7 | 8
score on a scale
  Week 4: number analyzed (Participants) | 5 | 7
  Week 4 | 22.2 (26.3) | 6 (11.3)
  Week 8 | 15.9 (26.3) | 6 (12.9)
  Week 12: number analyzed (Participants) | 3 | 6
  Week 12 | 44.7 (38.8) | 7.7 (18.3)

14. Secondary Outcome: 30-day Readmission Rate
Description: Percent of Group that was readmitted to the hospital within 30 days following hospital discharge.
Time Frame: 30 days from hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
Participants | 0 | 2

15. Secondary Outcome: Hospital Length of Stay (LOS)
Description: Hospital LOS was calculated from day of surgery to day of discharge from inpatient hospital ward to rehabilitation facility.
Time Frame: Number of days from surgery to discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
Number analyzed (Participants) | 8 | 8
days | 7 (1.6) | 6 (3.3)

ADVERSE EVENTS:
Time Frame: Week 4 and Week 8, Month 3, Month 6, and Month 12
Description: Subjects in the Control Group were not at risk for PNS Lead Reimplantation because they did not undergo implantation of any peripheral nerve stimulator leads. Other [Not Including Serious] Adverse Events were not monitored/assessed in the Control Arm/Group.
Arm/Group | Peripheral Nerve Stimulation (PNS) | Control
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Nerve Stimulation (PNS) (N=8) | Control (N=0)
PNS Lead Reimplantation (Surgical and medical procedures) | 2 (2) | 0 — Two subjects in the PNS group required reimplantation of PNS leads due to dislodgement. No suspected lead fractures were observed during the treatment period or lead removal.

LIMITATIONS AND CAVEATS:
Several participants underwent unanticipated amputation revisions, which has the potential to contribute to worsening pain and the need for increased opioids, which may significantly confound results. Subjects were instructed to use the device continuously, and the effects of PNS therapy may be impacted by the number of hours the device was utilized by the patient. Variations in subject compliance with device usage may impact outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT03484429/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03484429/ICF_001.pdf